CLINICAL TRIAL: NCT06043752
Title: Efficacy and Safety of Infliximab Biosimilar Remsima in Treatment of Chronic Plaque Psoriasis
Brief Title: Efficacy and Safety of Infliximab Biosimilar Remsima in Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ghurki Trust and Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — CT-P13

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remsima (Experimental)
  Interventions: Drug: Remsima

INTERVENTIONS:
Drug: Remsima — The patient will be given one Injection of REMSIMA 120 mg subcutaneously at week 0, 1, 2, 3, 4 and then every 2 weeks i.e., at 6, 8, 10 and 14 weeks. If the weight of the patient is >80 kg, 2 injections will be given.

SUMMARY:
Psoriasis is a persistent condition which demands prolonged management, so it puts heavy financial as well as psychological burden on patients. Severe psoriasis makes work impossible for patients. If it affects exposed parts of the body, it may lead to decrease in self-esteem, social avoidance, and shame. Patients with even mild form of psoriasis have high stigma as compared to other cutaneous diseases. As a result, psoriasis affected individuals experience greater difficulty in social interactions and employment. Patients experience symptoms in psoriasis includes bleeding, itching and inflamed joints. Psoriatic patients develop psoriatic arthritis approximately at 40 years of age which contributes to fatigue in these individuals. Moreover, early age onset of psoriasis leads to more physical impairment. Hence, patients get trapped in a vicious cycle as stress leads to further aggravation of disease. The European Medicine Agency has given its approval regarding the usage of INFLIXIMAB bio similar REMSIMA for psoriasis after taking in consideration its effectiveness from other studies conducted on ankylosing spondylitis and rheumatoid arthritis. This study is being conducted as no data is present on REMSIMA SC in psoriasis patient in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-59 years
* Both genders
* Diagnosed patient of Psoriasis
* Moderate to severe psoriasis
* Not responding to topical treatment
* Not responding to conventional systemic treatments i.e., methotrexate, cyclosporine and phototherapy.
* PASI score >10.

Exclusion Criteria:

Patient with active systemic lupus erythematosus or ANA positive patients.

* Patient with active tuberculosis.
* Extremely immunocompromised patient.
* Patient with cardiac disease.
* Patient with allergic reaction to REMSIMA.
* Pregnancy and Lactation.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area Severity Index Score | 24 weeks
  Patients will be followed 4,8,14 and 24 weeks
Adverse Events | 24 weeks
  Patients will be followed 4,8,14 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Haroon Nabi, Study Director — Professor Department of Dermatology LMDC; Dr. Nabigha Khalid, Principal Investigator — Department of Dermatology Ghurki Hospital; Dr. Saleha Batool, Study Chair — Assistant Professor Department of Dermatology, SIMS Hospital; Dr. Sumera Hanif, Study Chair — Senior Registrar Dermatology Department; Dr. Talat Masood Akbar, Study Chair — Associate Professor Dermatology LMDC GTTH; Dr. Faria Asad, Study Chair — Professor/ Head of Dermatology Department
Locations (1):
- Ghurki Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arsiwala S. Infliximab: efficacy in psoriasis. Indian J Dermatol Venereol Leprol. 2013 Jul;79 Suppl 7:S25-34. doi: 10.4103/0378-6323.115525. PMID 23974692
- [Background] Chaudhari U, Romano P, Mulcahy LD, Dooley LT, Baker DG, Gottlieb AB. Efficacy and safety of infliximab monotherapy for plaque-type psoriasis: a randomised trial. Lancet. 2001 Jun 9;357(9271):1842-7. doi: 10.1016/s0140-6736(00)04954-0. PMID 11410193
- [Background] Gisondi P, Bianchi L, Conti A, Dapavo P, Malagoli P, Piaserico S, Savoia F, Prignano F, Girolomoni G. Infliximab biosimilar CT-P13 in the treatment of chronic plaque psoriasis: data from the Psobiosimilars registry. Br J Dermatol. 2017 Dec;177(6):e325-e326. doi: 10.1111/bjd.15659. Epub 2017 Nov 22. No abstract available. PMID 28498543